CLINICAL TRIAL: NCT01656525
Title: A Multi-center, Multiple-ascending Dose, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability and Pharmacokinetics of Gantenerumab Following Subcutaneous Injection in Japanese AD Patients
Brief Title: A Multiple-dose Study of Gantenerumab in Japanese Alzheimer&Apos;s Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JP22431; JapicCTI-121849 (Registry Identifier: JAPIC)
Record Dates: First submitted 2012-06-05; First posted 2012-08-03 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Gantenerumab
- 2 (Experimental)
  Interventions: Drug: Gantenerumab
- 3 (Experimental)
  Interventions: Drug: Gantenerumab
- 4 (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gantenerumab — 75 mg subcutaneous doses every 4 weeks for 24 weeks
  Arms: 1
Drug: Gantenerumab — 105 mg subcutaneous doses every 4 weeks for 24 weeks
  Arms: 2
Drug: Gantenerumab — 225 mg subcutaneous doses every 4 weeks for 24 weeks
  Arms: 3
Drug: Placebo — subcutaneous doses every 4 weeks for 24 weeks
  Arms: 4

SUMMARY:
Objective of this study is to evaluate the safety, tolerability, pharmacokinetics and preliminary pharmacodynamic effects of multiple doses of Gantenerumab in subject with mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of probable AD dementia, based on NINCDS/ADRDA criteria
* Meet DSM-IV criteria for Dementia of the Alzheimer type
* MMSE score : 16 to 26 etc.

Exclusion Criteria:

* Meet the exclusion criteria of MRI at screening.
* A history of significant neurodegenerative diseases or dementia other than Alzheimer's disease.

etc.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 36 weeks
Pharmacokinetic parameters of Gantenerumab in plasma | 36 weeks
CSF/plasma ratios of Gantenerumab. | Baseline, Day183

SECONDARY OUTCOMES:
Change from baseline in plasma Abeta | Baseline,Day183
Change from baseline in plasma and CSF tau | Baseline,Day183
Change from baseline in Mini-Mental State Examination (MMSE) and Alzheimer's disease assessment scale cognitive behaviors (ADAS-Cog). | Baseline,Day85, 197, 253

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Kansai region, Kansai
  - Kanto region,, Kanto
  - Kyushu region, Kyushu
  - Tokai region, Toakai
  - Tohoku region, Tōhoku